CLINICAL TRIAL: NCT02906462
Title: Impact of an Early and Collegial Consideration of Patients' Vulnerability Comparing to Usual Care. Cluster Randomized Control Study "Mort-A-l'Hôpital 2"
Brief Title: Impact of an Early Palliative Approach
Acronym: MAHO2
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Investigator's decision (departure from institution)
Sponsor: Hopital Foch (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2013/99; 2012-A00444-39 (Other: ANSM)
Record Dates: First submitted 2016-02-17; First posted 2016-09-20 (Estimated); Last update posted 2019-05-17 (Actual); Status verified 2019-05

CONDITIONS: Incurable Disease
Keywords: Leonetti French law; Palliative care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual Practices (Other): Usual Practices
  Interventions: Other: Usual practices
- Early consideration of vulnerability (Other): Strategy promoting early consideration of patients' vulnerability
  Interventions: Other: Early consideration of vulnerability

INTERVENTIONS:
Other: Early consideration of vulnerability — One day training with the provision of vulnerability criteria inciting an early reflection of the level of therapeutic engagement; sheets available on the internet computer support collegial reflection and traceability of decisions to limit and stop treatments, incorporating the provisions of law known Leonetti
  Arms: Early consideration of vulnerability
Other: Usual practices — the centres applies their usual practices
  Arms: Usual Practices

SUMMARY:
In 2003, MAHO study (Ferrand E, Jabre P, Vincent-Genod C, et al. Circumstances of death in hospitalized patients and nurses' perceptions: French multicenter Mort-a-l'Hôpital survey. Arch Intern Med. 2008 168: 867-875.) evaluated the way 3793 patients died in 200 French hospitals and showed that their conditions of death were not optimal. The 22th April 2005 French Law precised patient's end of life rights with necessity to refrain from any unreasonable obstinacy, the right to refuse treatments and the obligation of a collegial process decision when the patient is not conscious. Since then, studies haven't demonstrate any improvement and found that palliative strategy in France is much less used than in other developed countries.

DETAILED DESCRIPTION:
In 2003, MAHO study evaluated the way 3793 patients died en 200 French hospitals and showed that their conditions of death were not optimal. The 22th April 2005 French Law precised patient's end of life rights with necessity to refrain from any unreasonable obstinacy, the right to refuse treatments and the obligation of a collegial process decision when the patient is not conscious. Since then, studies haven't demonstrate any improvement and found that palliative strategy in France is much less used than in other developed countries.

Principal Objective: To evaluate the impact of an early palliative strategy using vulnerability criteria compared to standard care.

Primary endpoint: Rate of withdraw/withhold of treatment in each group.

Secondary objectives: To evaluate the impact of early recognition of patients' vulnerability on death conditions ; to evaluate this strategy impact according to unit type on length of stay, palliative strategy modalities and caregivers' satisfaction.

Secondary endpoints: Rate of therapeutic involvement reflections ; rate of death following withholding or withdrawing of treatments ; traceability of the level of therapeutic involvement process ; Rate of patients deceased with their relatives next to them ; rate of patients deceased with comfort treatment ; rate of palliative care consultation before death ; rate of asks for euthanasia ; Doctor and nurse's perception of quality of support and death process of the patient

Methods: Prospective, controlled, cluster randomized study of routine care 2 groups:

* Group A: standard care and practice after 1 day of training
* Group B: 1 day of training, learning the vulnerability criteria that should induce early thinking about level of therapeutic involvement; web accessed forms will be available to help collegial process, withhold and withdraw decisions traceability, using legal requirements Number of patients to include: To detect a 20% absolute difference in palliative strategy used (30 to 50%), we determined that 5040 patients would provide a power of 80% with the use of a two-sided alpha level of 0.05. Sequential analysis is planned in order to early stop the study in case of efficacy or futility (minimal inclusion: 500 patients)

Inclusion criteria:

All patients hospitalized with at least one of the following vulnerability criteria will be included:

* Evolutive and symptomatic incurable cancer
* Aged more than 75 years old and presenting several geriatric syndromes (cognitive disorders, isolation, malnutrition, bedridden more than 12h per day)
* Neurologic pathology, chronic, with loss of autonomy (Performance Status>3)
* Final organ failure (heart, lungs, liver, kidney) with loss of autonomy (Performance Status>3)
* Care refusal and/or expressed will to die or repeated request for help to die

Exclusion criteria:

* Minors
* Patients without indication for treatment or surveillance with length of stay inferior to 24h
* Brain dead patients
* Not consent patients

Duration: 37 months (28 inclusion months for each center and a follow-up to hospital discharge, death or 9 months if the patient is still hospitalized).

Number of participating centers: 20 centers (28 services) were selected and recruit after training program among centers that did not used a formalized process to initiate level of therapeutic involvement reflection.

ELIGIBILITY:
Inclusion Criteria:

* Patient more than 18 years old hospitalized for at least 24h and who's prognosis (survival or quality of life) should lead to a palliative approach
* Patient suffering with at least one of the following vulnerability criteria will be included:

  * Evolutive and symptomatic incurable cancer
  * Aged more than 75 years old and presenting several geriatric syndromes (cognitive disorders, isolation, malnutrition, bedridden more than 12h per day)
  * Neurologic pathology, chronic, with loss of autonomy (Performance Status>3)
  * Final organ failure (heart, lungs, liver, kidney) with loss of autonomy (Performance Status>3)
  * Care refusal and/or expressed will to die or repeated request for help to die
* No opposition to the use of data collected from the patient or a relative or inclusion in emergency and non-opposition collected offline

Exclusion Criteria:

* Minors
* Patients without indication for treatment or surveillance with length of stay inferior to 24h
* Brain dead patients
* Not consent patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1200 (Estimated)
Dates: Start 2013-11; Primary Completion 2019-03 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
Rate of withdraw/withhold of treatment in each group | From hospital admission to death or discharge or 9 months after inclusion if the patient is still in the hospital
  To evaluate the impact of an early palliative strategy using vulnerability criteria compared to standard care.

SECONDARY OUTCOMES:
Death conditions | From hospital admission to death or discharge or 9 months after inclusion if the patient is still in the hospital
  rate of death relied to a withholding/withdrawing treatment decision, rate relatives present at the time of death, rate of death with comfort drugs, rate of patient/family/relatives interview with a psychologist.
  rate of death relied to a withholding/withdrawing treatment decision, rate relatives present at the time of death, rate of death with comfort drugs, rate of patient/family/relatives interview with a psychologist.
Early vulnerability consideration impact on length of stay | From hospital admission to death or discharge or 9 months after inclusion if the patient is still in the hospital
  total length of stay in the hospital
Palliative strategy modalities | From hospital admission to death or discharge or 9 months after inclusion if the patient is still in the hospital
  rate of reflections on level of therapeutic involvement
Early vulnerability consideration impact on caregivers' satisfaction | From hospital admission to death or discharge or 9 months after inclusion if the patient is still in the hospital
  Physician and nurses' perceptions about care management and conditions of death, caregivers interview with a psychologist

CONTACTS AND LOCATIONS:
Overall Officials: Edouard Ferrand, MD, Principal Investigator — e.ferrand@hopital-foch.org
Locations (23):
- France (23):
  - CHU, Amiens
  - Hopital privé Oncologie Médicale, Antony
  - Hôpital Privé Medecine interne, Antony
  - Hôpital Avicenne, Bobigny
  - Hôpital Ambroise Paré, Boulogne-Billancourt
  - Hôpital Georges Clemenceau, Champcueil
  - CHU, Dijon
  - Centre Hospitalier, Épernay
  - Hôpital Bicêtre, Le Kremlin-Bicêtre
  - CHRU, Lille
  - Hopital Lariboisiere Medecine interne, Paris
  - Groupe Hospitalier Paris - Saint-Joseph, Paris
  - Hopital Cochin Gastro-Enterologie, Paris
  - Centre Hospitalier Universitaire, Poitiers
  - Centre Hospitalier, Roubaix
  - Centre Hospitalier de Soissons, Soissons
  - Hiopital Foch Néphrologie, Suresnes
  - Hopital Foch Cardiologie, Suresnes
  - Hopital Foch Chirurgie Urologique, Suresnes
  - Hopital Foch Médecine Interne, Suresnes
  - Hopital Foch Neurochirurgie, Suresnes
  - Hopîtal Foch Urgences, Suresnes
  - CH, Valenciennes

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Truog RD, Cist AF, Brackett SE, Burns JP, Curley MA, Danis M, DeVita MA, Rosenbaum SH, Rothenberg DM, Sprung CL, Webb SA, Wlody GS, Hurford WE. Recommendations for end-of-life care in the intensive care unit: The Ethics Committee of the Society of Critical Care Medicine. Crit Care Med. 2001 Dec;29(12):2332-48. doi: 10.1097/00003246-200112000-00017. No abstract available. PMID 11801837
- [Result] Ferrand E, Jabre P, Vincent-Genod C, Aubry R, Badet M, Badia P, Cariou A, Ellien F, Gounant V, Gil R, Jaber S, Jay S, Paillaud E, Poulain P, Regnier B, Reignier J, Socie G, Tardy B, Lemaire F, Brun-Buisson C, Marty J; French Mort-a-l'Hopital Group. Circumstances of death in hospitalized patients and nurses' perceptions: French multicenter Mort-a-l'Hopital survey. Arch Intern Med. 2008 Apr 28;168(8):867-75. doi: 10.1001/archinte.168.8.867. PMID 18443263
- [Result] Ferrand E, Robert R, Ingrand P, Lemaire F; French LATAREA Group. Withholding and withdrawal of life support in intensive-care units in France: a prospective survey. French LATAREA Group. Lancet. 2001 Jan 6;357(9249):9-14. doi: 10.1016/s0140-6736(00)03564-9. PMID 11197395
- [Result] Ferrand E, Lemaire F, Regnier B, Kuteifan K, Badet M, Asfar P, Jaber S, Chagnon JL, Renault A, Robert R, Pochard F, Herve C, Brun-Buisson C, Duvaldestin P; French RESSENTI Group. Discrepancies between perceptions by physicians and nursing staff of intensive care unit end-of-life decisions. Am J Respir Crit Care Med. 2003 May 15;167(10):1310-5. doi: 10.1164/rccm.200207-752OC. Epub 2003 Jan 24. PMID 12738597
- [Result] Ferrand E, Marty J; French LATASAMU Group. Prehospital withholding and withdrawal of life-sustaining treatments. The French LATASAMU survey. Intensive Care Med. 2006 Oct;32(10):1498-505. doi: 10.1007/s00134-006-0292-5. Epub 2006 Aug 2. PMID 16896861
- [Result] Prendergast TJ, Claessens MT, Luce JM. A national survey of end-of-life care for critically ill patients. Am J Respir Crit Care Med. 1998 Oct;158(4):1163-7. doi: 10.1164/ajrccm.158.4.9801108. PMID 9769276
- [Result] Sprung CL, Cohen SL, Sjokvist P, Baras M, Bulow HH, Hovilehto S, Ledoux D, Lippert A, Maia P, Phelan D, Schobersberger W, Wennberg E, Woodcock T; Ethicus Study Group. End-of-life practices in European intensive care units: the Ethicus Study. JAMA. 2003 Aug 13;290(6):790-7. doi: 10.1001/jama.290.6.790. PMID 12915432
- [Result] Ferrand E, Jabre P, Fernandez-Curiel S, Morin F, Vincent-Genod C, Duvaldestin P, Lemaire F, Herve C, Marty J. Participation of French general practitioners in end-of-life decisions for their hospitalised patients. J Med Ethics. 2006 Dec;32(12):683-7. doi: 10.1136/jme.2005.014084. PMID 17145904
- [Result] Temel JS, Greer JA, Muzikansky A, Gallagher ER, Admane S, Jackson VA, Dahlin CM, Blinderman CD, Jacobsen J, Pirl WF, Billings JA, Lynch TJ. Early palliative care for patients with metastatic non-small-cell lung cancer. N Engl J Med. 2010 Aug 19;363(8):733-42. doi: 10.1056/NEJMoa1000678. PMID 20818875
- [Result] Kelley AS, Meier DE. Palliative care--a shifting paradigm. N Engl J Med. 2010 Aug 19;363(8):781-2. doi: 10.1056/NEJMe1004139. No abstract available. PMID 20818881
- [Result] Greer JA, Pirl WF, Jackson VA, Muzikansky A, Lennes IT, Heist RS, Gallagher ER, Temel JS. Effect of early palliative care on chemotherapy use and end-of-life care in patients with metastatic non-small-cell lung cancer. J Clin Oncol. 2012 Feb 1;30(4):394-400. doi: 10.1200/JCO.2011.35.7996. Epub 2011 Dec 27. PMID 22203758
- [Result] Yoong J, Park ER, Greer JA, Jackson VA, Gallagher ER, Pirl WF, Back AL, Temel JS. Early palliative care in advanced lung cancer: a qualitative study. JAMA Intern Med. 2013 Feb 25;173(4):283-90. doi: 10.1001/jamainternmed.2013.1874. PMID 23358690